CLINICAL TRIAL: NCT06056791
Title: An Open-label, Phase I/IIa Dose Escalation and Expansion Study to Determine the Safety and Clinical Activity of an Immune Priming Cell Therapy (INKmune) in Patients With Metastatic Castration Resistant Prostate Cancer (mCRPC)
Brief Title: Study of INKmune in Patients With mCRPC (CaRe Prostate)
Acronym: CaRe
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Inmune Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INMB-INB16-003
Record Dates: First submitted 2023-08-07; First posted 2023-09-28 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Metastatic Castration-resistant Prostate Cancer; mCRPC
Keywords: mCRPC; NK Cell Based Therapy; Immune Mediated Therapy; Cell Therapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Dose escalation using mBOIN design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1: 1 x 10^8 INKmune (Experimental): In Dose Escalation: INKmune therapy will be administered by a slow intravenous injection via conventional blood giving set. Approximately 18 patients will receive 3 weekly IV doses of INKmune on Day 1, 8, and 15 as per the below:
  * In Cohort 1, the initial planned dose is 1 x 10^8 INKmune;
  * In Cohort 2, the weekly dose will increase to 3 x 10^8 INKmune;
  * In Cohort 3, the weekly dose will increase to 5 x 10^8 INKmune.
  In Dose Expansion: INKmune therapy will be administered by a slow intravenous injection via conventional blood giving set. Approximately 12 patients will receive 3 weekly IV doses of INKmune on Day 1, 8, and 15 as per the below:
  Following mBOIN termination and MTD identification, patients will be enrolled in up to two candidate optimal dose levels (no higher than the MTD) for final optimal dose determination.
  Interventions: Biological: INKmune
- Cohort 2: 3 x 10^8 INKmune (Experimental): In Dose Escalation: INKmune therapy will be administered by a slow intravenous injection via conventional blood giving set. Approximately 18 patients will receive 3 weekly IV doses of INKmune on Day 1, 8, and 15 as per the below:
  * In Cohort 1, the initial planned dose is 1 x 10^8 INKmune;
  * In Cohort 2, the weekly dose will increase to 3 x 10^8 INKmune;
  * In Cohort 3, the weekly dose will increase to 5 x 10^8 INKmune.
  In Dose Expansion: INKmune therapy will be administered by a slow intravenous injection via conventional blood giving set. Approximately 12 patients will receive 3 weekly IV doses of INKmune on Day 1, 8, and 15 as per the below:
  Following mBOIN termination and MTD identification, patients will be enrolled in up to two candidate optimal dose levels (no higher than the MTD) for final optimal dose determination.
  Interventions: Biological: INKmune
- Cohort 3: 5 x 10^8 INKmune (Experimental): In Dose Escalation: INKmune therapy will be administered by a slow intravenous injection via conventional blood giving set. Approximately 18 patients will receive 3 weekly IV doses of INKmune on Day 1, 8, and 15 as per the below:
  * In Cohort 1, the initial planned dose is 1 x 10^8 INKmune;
  * In Cohort 2, the weekly dose will increase to 3 x 10^8 INKmune;
  * In Cohort 3, the weekly dose will increase to 5 x 10^8 INKmune.
  In Dose Expansion: INKmune therapy will be administered by a slow intravenous injection via conventional blood giving set. Approximately 12 patients will receive 3 weekly IV doses of INKmune on Day 1, 8, and 15 as per the below:
  Following mBOIN termination and MTD identification, patients will be enrolled in up to two candidate optimal dose levels (no higher than the MTD) for final optimal dose determination.
  Interventions: Biological: INKmune

INTERVENTIONS:
Biological: INKmune — INKmune is a patented biologic delivery system and method for cancer treatment using in vivo priming and activation of natural killer (NK) cells in order to achieve tumor cell lysis. INKmune is a suspension of INB16 cells which have been rendered replication incompetent that does not require donor matching.

SUMMARY:
This is an open-label, phase I/IIa dose escalation and expansion study of INKmune in men with mCRPC. INKmune is administered to patients intravenously over three doses, at least one-week apart. The study will consist of two stages.

DETAILED DESCRIPTION:
This is an open-label, phase I/IIa dose escalation and expansion study of INKmune in men with mCRPC. INKmune is administered to patients intravenously over 3 doses. The 3 infusions will occur over a minimum of a 2-week period, with each infusion at least 1 week apart. The study will consist of 2 stages:

* Dose escalation: exploring dose levels of 1x10^8, 3x10^8, and 5x10^8 cells per infusion.
* Dose expansion: following mBOIN termination and maximum tolerated dose (MTD) identification, patients will be enrolled in up to 2 candidate optimal dose levels for final optimal dose determination.

Eligible patients will sign informed consent prior to any study assessments being performed. Patients have up to 30 days in which to have all screening procedures and eligibility assessed. Patients will be infused with INKmune on Days 1, 8, and 15. Patients will also present to site on days 29, 57, 85, 113, and 141 to complete study assessments. Day 169 is the last study visit and patient will have completed trial after this visit has been completed. Option to enroll in the INKmune Long term Follow-up Registry will be presented at Day 169 visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects over 18 years of age at time of screening.
2. Blood Prostate Specific Antigen (PSA) of >1.0 ng/ml at time of screening.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1 at time of screening.
4. Histologic confirmation of adenocarcinoma prostate cancer.
5. A diagnosis of progressive metastatic castrate resistant prostate cancer (mCRPC), as defined by Prostate Cancer Clinical Trials Working Group 3 (PCWG3), following androgen deprivation therapy (ADT) and at least one androgen receptor signaling inhibitor, but not more than 3 therapies in addition to ADT. Progressive disease at the time of study entry as indicated by at least one of the following:

   * i. At least two rising PSA values at a minimum of a one-week interval. If PSA is the only measure of progression, then the minimum PSA value at the start of treatment must be ≥ 1 ng/mL.
   * ii. Radiographic progression per RECIST1.1 for soft tissue (at least 1 measurable lesion per RECIST 1.1), and/or
   * iii. Progression of bone metastases.
6. Castrate level of testosterone of < 50 ng/dL.
7. Adequate organ function indicated by the following laboratory parameters:

   * i. Hemoglobin ≥ 8.0 g/dL.
   * ii. White Blood Cell Count (WBC) ≥ 3.0 x 10⁹/L.
   * iii. Lymphocytes ≥ 80% LLN
   * iv. Absolute Neutrophil Count (ANC) ≥ 1.5 x 10⁹/L.
   * v. Platelets ≥ 100 x 10⁹/L.
   * vi. PT and APTT < 1.5x ULN (unless receiving therapeutic anticoagulation).
   * vii. AST or ALT ≤ 2.5x ULN. AST or ALT ≤ 5x ULN for patients with liver metastases.
   * viii. Bilirubin < 1.5x ULN (< 3x ULN in Gilbert's Syndrome).
   * ix. Creatinine clearance/estimated GFR ≥ 30 mL/min (MDRD or Cockcroft-Gault).
   * x. Resting room air PaO2 saturation of >95% as measured by pulse oximetry.
8. Negative screen for Human Immunodeficiency virus (HIV), Hepatitis B virus (HBV) antigen, and Hepatitis C virus (HCV). If testing was done within the past three months, there is no need to repeat testing if documentation of results is provided to the study site.
9. Subjects and their partners of reproductive potential must agree to use an effective form of contraception during the period of drug administration and for three months following the completion of the last administration of the study drug. An effective form of contraception is defined as oral contraceptives plus one form of barrier method or double barrier methods (condom with spermicide or condom with diaphragm).
10. Subjects must be able to understand the potential risks and benefits of the study and be able to read and give written informed consent.

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

1. Diagnosis of small cell/neuroendocrine prostate cancer. Immunohistochemical staining for neuroendocrine markers (e.g., chromogranin A, neuron-specific enolase, and synaptophysin) is not sufficient to establish a small cell/neuroendocrine histology; morphologic features that are characteristic of small cell/neuroendocrine prostate cancer are required to confirm the presence of small cell/neuroendocrine prostate cancer.
2. History of concurrent malignant cancer within previous 3 years, with the exception of in situ carcinomas and non-melanoma skin cancer. If diagnosis or treatment for other cancers have occurred in the last 3 years, further discussion needed.
3. Uncontrolled autoimmune disease including, but not limited to, systemic lupus erythematosus, rheumatoid arthritis, ulcerative colitis, Crohn's disease, temporal arteritis, and thyroiditis. Autoimmune conditions that are well-controlled in the opinion of the investigator must first be discussed with the Sponsor prior to enrollment.
4. A requirement for daily systemic corticosteroids for any reason; or other immunosuppressive or immunomodulatory agents. Topical, nasal, modified-release oral, and/or physiologic corticosteroids may be permitted following discussion with the Sponsor.
5. Clinically significant cardiac disease (New York Heart Association Class III/IV) or severe debilitating pulmonary disease.
6. Patients with a current or recent history, as determined by the Investigator, of clinically significant, progressive, and/or uncontrolled renal, hepatic, hematological, endocrine, pulmonary, cardiac, gastroenterological, or neurological disease.
7. Cytotoxic chemotherapy within three weeks prior to start of study treatment (Day 1).
8. Radiation therapy within two weeks prior to start of study treatment (Day 1).
9. Patients may not have received a previous NK based therapy.
10. Evidence of central nervous system (CNS) metastatic disease at screening.
11. Patients with an active infection requiring antibiotic treatment within seven days of starting study treatment (Day 1).
12. Administration of live attenuated vaccines within eight weeks of start of study treatment (Day 1) and throughout the study.
13. Any other medical condition that in the opinion of the Investigator may interfere with a subject's participation in, or compliance with, the study
14. Participation in a therapeutic research study or receipt of an investigational drug within 4 weeks of start of treatment (Day 1) or 5 half-lives, whichever occurs first.
15. Expected survival of less than six months
16. At the time of consent, unable to comply with study procedures and assessments.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Determine the optimal concentration of INKmune therapy to be used in patients with mCRPC. | 2-3 years
  Measurement of peripheral blood activated NK cell (memory like NK cell phenotype) percentage by flow cytometry to >2 times pre-treatment percentage.
Determine the optimal concentration of INKmune therapy to be used in patients with mCRPC. | 2-3 years
  Measurement of Prostate Specific Antigen (PSA) to determine the percent of patients that decrease PSA by ≥30% during treatment.
Determine the optimal concentration of INKmune therapy to be used in patients with mCRPC. | 2-3 years
  Measurement of disease burden as determined by prostate-specific membrane antigen (PMSA) positron emission tomography (PET) scan.
Determine the optimal concentration of INKmune therapy to be used in patients with mCRPC. | 2-3 years
  Measurement of change in circulating tumor DNA (ctDNA).
Evaluate the safety and tolerability of INKmune therapy in patients with mCRPC. | 2-3 years
  Measurement of frequency and severity of Dose-Limiting Toxicities (DLT).
Evaluate the safety and tolerability of INKmune therapy in patients with mCRPC. | 2-3 years
  MTD identification, if available.
Evaluate the safety and tolerability of INKmune therapy in patients with mCRPC. | 2-3 years
  Measurement of frequency and severity of adverse events (AEs).
Evaluate the safety and tolerability of INKmune therapy in patients with mCRPC. | 2-3 years
  Measurement of frequency and severity of serious adverse events (SAEs).

SECONDARY OUTCOMES:
Evaluate the overall clinical efficacy of INKmune treatment in patients utilizing RECIST. | 2-3 years
  Assessment based on current Prostate Cancer Working Group 3 (PCWG3) modified Response Evaluation Criteria (RECIST) Version 1.1, where applicable.
Evaluate the overall clinical efficacy of INKmune treatment in patients utilizing PSA. | 2-3 years
  Measurement of PSA response using PSA50 response rate.
Evaluate the overall clinical efficacy of INKmune treatment in patients utilizing PSA. | 2-3 years
  Measurement of the period of time PSA decrease by ≥30%.
Evaluate the overall clinical efficacy of INKmune treatment in patients utilizing PSA. | 2-3 years
  Measurement of the period of time PSA is below baseline.
Evaluate the overall clinical efficacy of INKmune treatment in patients utilizing survival data. | 2-3 years
  Measurement of Progression Free Survival (PFS).
Evaluate the overall clinical efficacy of INKmune treatment in patients utilizing survival data. | 2-3 years
  Measurement of Radiological Progression Free Survival (rPFS).
Evaluate the overall clinical efficacy of INKmune treatment in patients utilizing disease response. | 2-3 years
  Measurement of Objective response rate (ORR)
Evaluate the overall clinical efficacy of INKmune treatment in patients utilizing disease response. | 2-3 years
  Measurement of the Disease control rate.
Evaluate the overall clinical efficacy of INKmune treatment in patients utilizing survival data. | 2-3 years
  Measurement of Overall survival (OS).

OTHER OUTCOMES:
Assess persistence of memory like Natural Killer (NK) cell number. | 2-3 years
  Assess persistence of memory like Natural Killer (NK) cell number.
Explore the relationship between persistence of INKmune cells in patients treated with INKmune and disease response experienced through Day 169. | 1-169 Days
  Relationship will be explored through multi-parameter flow cytometry and tumor killing of NK resistant tumor targets (RAJI cells) in blood of patients after treatment with INKmune. Disease response will be assessed from RECIST, PSMA, PSA data.
Determine change in blood PSA levels compared to change in tumor burden, as assessed by RECIST v1.1, and Pylarify PSMA PET scan (piflufolastat F 18) for each patient treated with INKmune. | 1-169 Days
  Relationship between blood PSA levels and change in tumor burden will be assessed through collection of serum PSA level and measurable disease burden assessed by RECIST v1.1, PCWG3 criteria, and Pylarify PSMA PET scan (piflufolastat F 18). PSA will be collected at Screening and at each visit following the 3 doses of INKmune. PSMA PET scans will be completed at Day 1, Day 57 and Day 169.
Determine the concentration of circulating tumor DNA (ctDNA) levels and treatment response in patients with ctDNA data. | 1-169 Days
  Relationship between ctDNA levels and treatment response will be assessed by collection of serial ctDNA assays in patients with available pre-treatment tumor DNA. ctDNA collections will occur at Day 1, Day 57 and Day 169.
Determine endogenous NK cell infiltration from optional biopsy tissue and previously resected tissue (if available). | 2-3 years
  Optional biopsy tissue and previously resected tissue will be analyzed with Immunohistochemistry (IHC) and RNA sequencing of patient pathological specimens.
Determine stromal expression of inhibitory ligands from optional biopsy tissue and previously resected tissue (if available). | 2-3 years
  Optional biopsy tissue and previously resected tissue will be analyzed with Immunohistochemistry (IHC) and RNA sequencing of patient pathological specimens.
Complete transcriptomic analyses from optional biopsy tissue and previously resected tissue (if available). | 2-3 years
  Optional biopsy tissue and previously resected tissue will be analyzed with Immunohistochemistry (IHC) and RNA sequencing of patient pathological specimens.
Evaluate activity of INKmune therapy in relation to the sequence of mCRPC treatment received by patients. | 2-3 years
  Outcome will be evaluated by review of medical history and collection of safety follow-up visits to record mCRPC treatments after completion of clinical trial in comparison to peripheral blood activated NK cell (memory like NK cell phenotype) percentage by flow cytometry.
Assess the experience of clinical trial participation by patients through a comprehensive patient survey provided post visit at 3 timepoints during the trial. | 1-2 years
  Quality Improvement: Assess the experience of clinical trial participation by patients through patient questionnaires collected throughout the clinical trial. Questionnaires will be provided at 3 time points during study participation following study visits.
  Understand the patient experiences across participation in the clinical trial, through patient questionnaires (answers to be selected on a scale from '1 to 5', with '1' being very poor and '5' being very good), to assess patient perceptions in the following areas:
  * Access,
  * Communication,
  * Information & materials,
  * Patient burden,
  * Patient centeredness,
  * Privacy,
  * Quality of care,
  * Trust,
  * Safety.

CONTACTS AND LOCATIONS:
Overall Officials: Tara Lehner, Study Director — INmune Bio
Locations (8):
- United States (8):
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Carl & Edyth Lindner Center for Research and Education at The Christ Hospital and The Christ Hospital Cancer Center, Cincinnati, Ohio
  - Renovatio Clinical, El Paso, Texas
  - Renovatio Clinical, The Woodlands, Texas
  - NEXT Virginia, Fairfax, Virginia
  - VA Puget Sound Health Care System, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2018. CA Cancer J Clin. 2018 Jan;68(1):7-30. doi: 10.3322/caac.21442. Epub 2018 Jan 4. PMID 29313949
- [Background] Center MM, Jemal A, Lortet-Tieulent J, Ward E, Ferlay J, Brawley O, Bray F. International variation in prostate cancer incidence and mortality rates. Eur Urol. 2012 Jun;61(6):1079-92. doi: 10.1016/j.eururo.2012.02.054. Epub 2012 Mar 8. PMID 22424666
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Global Burden of Disease Cancer Collaboration; Fitzmaurice C, Akinyemiju TF, Al Lami FH, Alam T, Alizadeh-Navaei R, Allen C, Alsharif U, Alvis-Guzman N, Amini E, Anderson BO, Aremu O, Artaman A, Asgedom SW, Assadi R, Atey TM, Avila-Burgos L, Awasthi A, Ba Saleem HO, Barac A, Bennett JR, Bensenor IM, Bhakta N, Brenner H, Cahuana-Hurtado L, Castaneda-Orjuela CA, Catala-Lopez F, Choi JJ, Christopher DJ, Chung SC, Curado MP, Dandona L, Dandona R, das Neves J, Dey S, Dharmaratne SD, Doku DT, Driscoll TR, Dubey M, Ebrahimi H, Edessa D, El-Khatib Z, Endries AY, Fischer F, Force LM, Foreman KJ, Gebrehiwot SW, Gopalani SV, Grosso G, Gupta R, Gyawali B, Hamadeh RR, Hamidi S, Harvey J, Hassen HY, Hay RJ, Hay SI, Heibati B, Hiluf MK, Horita N, Hosgood HD, Ilesanmi OS, Innos K, Islami F, Jakovljevic MB, Johnson SC, Jonas JB, Kasaeian A, Kassa TD, Khader YS, Khan EA, Khan G, Khang YH, Khosravi MH, Khubchandani J, Kopec JA, Kumar GA, Kutz M, Lad DP, Lafranconi A, Lan Q, Legesse Y, Leigh J, Linn S, Lunevicius R, Majeed A, Malekzadeh R, Malta DC, Mantovani LG, McMahon BJ, Meier T, Melaku YA, Melku M, Memiah P, Mendoza W, Meretoja TJ, Mezgebe HB, Miller TR, Mohammed S, Mokdad AH, Moosazadeh M, Moraga P, Mousavi SM, Nangia V, Nguyen CT, Nong VM, Ogbo FA, Olagunju AT, Pa M, Park EK, Patel T, Pereira DM, Pishgar F, Postma MJ, Pourmalek F, Qorbani M, Rafay A, Rawaf S, Rawaf DL, Roshandel G, Safiri S, Salimzadeh H, Sanabria JR, Santric Milicevic MM, Sartorius B, Satpathy M, Sepanlou SG, Shackelford KA, Shaikh MA, Sharif-Alhoseini M, She J, Shin MJ, Shiue I, Shrime MG, Sinke AH, Sisay M, Sligar A, Sufiyan MB, Sykes BL, Tabares-Seisdedos R, Tessema GA, Topor-Madry R, Tran TT, Tran BX, Ukwaja KN, Vlassov VV, Vollset SE, Weiderpass E, Williams HC, Yimer NB, Yonemoto N, Younis MZ, Murray CJL, Naghavi M. Global, Regional, and National Cancer Incidence, Mortality, Years of Life Lost, Years Lived With Disability, and Disability-Adjusted Life-Years for 29 Cancer Groups, 1990 to 2016: A Systematic Analysis for the Global Burden of Disease Study. JAMA Oncol. 2018 Nov 1;4(11):1553-1568. doi: 10.1001/jamaoncol.2018.2706. PMID 29860482
- [Background] Negoita S, Feuer EJ, Mariotto A, Cronin KA, Petkov VI, Hussey SK, Benard V, Henley SJ, Anderson RN, Fedewa S, Sherman RL, Kohler BA, Dearmon BJ, Lake AJ, Ma J, Richardson LC, Jemal A, Penberthy L. Annual Report to the Nation on the Status of Cancer, part II: Recent changes in prostate cancer trends and disease characteristics. Cancer. 2018 Jul 1;124(13):2801-2814. doi: 10.1002/cncr.31549. Epub 2018 May 22. PMID 29786851
- [Background] Flaig TW, Potluri RC, Ng Y, Todd MB, Mehra M. Treatment evolution for metastatic castration-resistant prostate cancer with recent introduction of novel agents: retrospective analysis of real-world data. Cancer Med. 2016 Feb;5(2):182-91. doi: 10.1002/cam4.576. Epub 2015 Dec 29. PMID 26710718
- [Background] Beer TM, Armstrong AJ, Rathkopf DE, Loriot Y, Sternberg CN, Higano CS, Iversen P, Bhattacharya S, Carles J, Chowdhury S, Davis ID, de Bono JS, Evans CP, Fizazi K, Joshua AM, Kim CS, Kimura G, Mainwaring P, Mansbach H, Miller K, Noonberg SB, Perabo F, Phung D, Saad F, Scher HI, Taplin ME, Venner PM, Tombal B; PREVAIL Investigators. Enzalutamide in metastatic prostate cancer before chemotherapy. N Engl J Med. 2014 Jul 31;371(5):424-33. doi: 10.1056/NEJMoa1405095. Epub 2014 Jun 1. PMID 24881730
- [Background] Ryan CJ, Smith MR, de Bono JS, Molina A, Logothetis CJ, de Souza P, Fizazi K, Mainwaring P, Piulats JM, Ng S, Carles J, Mulders PF, Basch E, Small EJ, Saad F, Schrijvers D, Van Poppel H, Mukherjee SD, Suttmann H, Gerritsen WR, Flaig TW, George DJ, Yu EY, Efstathiou E, Pantuck A, Winquist E, Higano CS, Taplin ME, Park Y, Kheoh T, Griffin T, Scher HI, Rathkopf DE; COU-AA-302 Investigators. Abiraterone in metastatic prostate cancer without previous chemotherapy. N Engl J Med. 2013 Jan 10;368(2):138-48. doi: 10.1056/NEJMoa1209096. Epub 2012 Dec 10. PMID 23228172
- [Background] Cheng HH, Gulati R, Azad A, Nadal R, Twardowski P, Vaishampayan UN, Agarwal N, Heath EI, Pal SK, Rehman HT, Leiter A, Batten JA, Montgomery RB, Galsky MD, Antonarakis ES, Chi KN, Yu EY. Activity of enzalutamide in men with metastatic castration-resistant prostate cancer is affected by prior treatment with abiraterone and/or docetaxel. Prostate Cancer Prostatic Dis. 2015 Jun;18(2):122-7. doi: 10.1038/pcan.2014.53. Epub 2015 Jan 20. PMID 25600186
- [Background] Suzman DL, Luber B, Schweizer MT, Nadal R, Antonarakis ES. Clinical activity of enzalutamide versus docetaxel in men with castration-resistant prostate cancer progressing after abiraterone. Prostate. 2014 Sep;74(13):1278-85. doi: 10.1002/pros.22844. Epub 2014 Jul 22. PMID 25053178
- [Background] Tannock IF, de Wit R, Berry WR, Horti J, Pluzanska A, Chi KN, Oudard S, Theodore C, James ND, Turesson I, Rosenthal MA, Eisenberger MA; TAX 327 Investigators. Docetaxel plus prednisone or mitoxantrone plus prednisone for advanced prostate cancer. N Engl J Med. 2004 Oct 7;351(15):1502-12. doi: 10.1056/NEJMoa040720. PMID 15470213
- [Background] de Bono JS, Oudard S, Ozguroglu M, Hansen S, Machiels JP, Kocak I, Gravis G, Bodrogi I, Mackenzie MJ, Shen L, Roessner M, Gupta S, Sartor AO; TROPIC Investigators. Prednisone plus cabazitaxel or mitoxantrone for metastatic castration-resistant prostate cancer progressing after docetaxel treatment: a randomised open-label trial. Lancet. 2010 Oct 2;376(9747):1147-54. doi: 10.1016/S0140-6736(10)61389-X. PMID 20888992
- [Background] Crawford ED, Higano CS, Shore ND, Hussain M, Petrylak DP. Treating Patients with Metastatic Castration Resistant Prostate Cancer: A Comprehensive Review of Available Therapies. J Urol. 2015 Dec;194(6):1537-47. doi: 10.1016/j.juro.2015.06.106. Epub 2015 Jul 18. PMID 26196735
- [Background] Gray PJ, Lin CC, Cooperberg MR, Jemal A, Efstathiou JA. Temporal Trends and the Impact of Race, Insurance, and Socioeconomic Status in the Management of Localized Prostate Cancer. Eur Urol. 2017 May;71(5):729-737. doi: 10.1016/j.eururo.2016.08.047. Epub 2016 Sep 3. PMID 27597241
- [Background] Loeb S, Bruinsma SM, Nicholson J, Briganti A, Pickles T, Kakehi Y, Carlsson SV, Roobol MJ. Active surveillance for prostate cancer: a systematic review of clinicopathologic variables and biomarkers for risk stratification. Eur Urol. 2015 Apr;67(4):619-26. doi: 10.1016/j.eururo.2014.10.010. Epub 2014 Oct 31. PMID 25457014
- [Background] Resnick MJ, Koyama T, Fan KH, Albertsen PC, Goodman M, Hamilton AS, Hoffman RM, Potosky AL, Stanford JL, Stroup AM, Van Horn RL, Penson DF. Long-term functional outcomes after treatment for localized prostate cancer. N Engl J Med. 2013 Jan 31;368(5):436-45. doi: 10.1056/NEJMoa1209978. PMID 23363497
- [Background] Vlachostergios PJ, Puca L, Beltran H. Emerging Variants of Castration-Resistant Prostate Cancer. Curr Oncol Rep. 2017 May;19(5):32. doi: 10.1007/s11912-017-0593-6. PMID 28361223
- [Background] Knudsen KE, Penning TM. Partners in crime: deregulation of AR activity and androgen synthesis in prostate cancer. Trends Endocrinol Metab. 2010 May;21(5):315-24. doi: 10.1016/j.tem.2010.01.002. Epub 2010 Feb 6. PMID 20138542
- [Background] James ND, Sydes MR, Clarke NW, Mason MD, Dearnaley DP, Spears MR, Ritchie AW, Parker CC, Russell JM, Attard G, de Bono J, Cross W, Jones RJ, Thalmann G, Amos C, Matheson D, Millman R, Alzouebi M, Beesley S, Birtle AJ, Brock S, Cathomas R, Chakraborti P, Chowdhury S, Cook A, Elliott T, Gale J, Gibbs S, Graham JD, Hetherington J, Hughes R, Laing R, McKinna F, McLaren DB, O'Sullivan JM, Parikh O, Peedell C, Protheroe A, Robinson AJ, Srihari N, Srinivasan R, Staffurth J, Sundar S, Tolan S, Tsang D, Wagstaff J, Parmar MK; STAMPEDE investigators. Addition of docetaxel, zoledronic acid, or both to first-line long-term hormone therapy in prostate cancer (STAMPEDE): survival results from an adaptive, multiarm, multistage, platform randomised controlled trial. Lancet. 2016 Mar 19;387(10024):1163-77. doi: 10.1016/S0140-6736(15)01037-5. Epub 2015 Dec 21. PMID 26719232
- [Background] Sweeney CJ, Chen YH, Carducci M, Liu G, Jarrard DF, Eisenberger M, Wong YN, Hahn N, Kohli M, Cooney MM, Dreicer R, Vogelzang NJ, Picus J, Shevrin D, Hussain M, Garcia JA, DiPaola RS. Chemohormonal Therapy in Metastatic Hormone-Sensitive Prostate Cancer. N Engl J Med. 2015 Aug 20;373(8):737-46. doi: 10.1056/NEJMoa1503747. Epub 2015 Aug 5. PMID 26244877
- [Background] Kyriakopoulos CE, Chen YH, Carducci MA, Liu G, Jarrard DF, Hahn NM, Shevrin DH, Dreicer R, Hussain M, Eisenberger M, Kohli M, Plimack ER, Vogelzang NJ, Picus J, Cooney MM, Garcia JA, DiPaola RS, Sweeney CJ. Chemohormonal Therapy in Metastatic Hormone-Sensitive Prostate Cancer: Long-Term Survival Analysis of the Randomized Phase III E3805 CHAARTED Trial. J Clin Oncol. 2018 Apr 10;36(11):1080-1087. doi: 10.1200/JCO.2017.75.3657. Epub 2018 Jan 31. PMID 29384722
- [Background] James ND, de Bono JS, Spears MR, Clarke NW, Mason MD, Dearnaley DP, Ritchie AWS, Amos CL, Gilson C, Jones RJ, Matheson D, Millman R, Attard G, Chowdhury S, Cross WR, Gillessen S, Parker CC, Russell JM, Berthold DR, Brawley C, Adab F, Aung S, Birtle AJ, Bowen J, Brock S, Chakraborti P, Ferguson C, Gale J, Gray E, Hingorani M, Hoskin PJ, Lester JF, Malik ZI, McKinna F, McPhail N, Money-Kyrle J, O'Sullivan J, Parikh O, Protheroe A, Robinson A, Srihari NN, Thomas C, Wagstaff J, Wylie J, Zarkar A, Parmar MKB, Sydes MR; STAMPEDE Investigators. Abiraterone for Prostate Cancer Not Previously Treated with Hormone Therapy. N Engl J Med. 2017 Jul 27;377(4):338-351. doi: 10.1056/NEJMoa1702900. Epub 2017 Jun 3. PMID 28578639
- [Background] Fizazi K, Tran N, Fein L, Matsubara N, Rodriguez-Antolin A, Alekseev BY, Ozguroglu M, Ye D, Feyerabend S, Protheroe A, De Porre P, Kheoh T, Park YC, Todd MB, Chi KN; LATITUDE Investigators. Abiraterone plus Prednisone in Metastatic, Castration-Sensitive Prostate Cancer. N Engl J Med. 2017 Jul 27;377(4):352-360. doi: 10.1056/NEJMoa1704174. Epub 2017 Jun 4. PMID 28578607
- [Background] Pezaro CJ, Omlin AG, Altavilla A, Lorente D, Ferraldeschi R, Bianchini D, Dearnaley D, Parker C, de Bono JS, Attard G. Activity of cabazitaxel in castration-resistant prostate cancer progressing after docetaxel and next-generation endocrine agents. Eur Urol. 2014 Sep;66(3):459-65. doi: 10.1016/j.eururo.2013.11.044. Epub 2013 Dec 17. PMID 24411987
- [Background] Handy CE, Antonarakis ES. Sequencing Treatment for Castration-Resistant Prostate Cancer. Curr Treat Options Oncol. 2016 Dec;17(12):64. doi: 10.1007/s11864-016-0438-9. PMID 27822685
- [Background] Zhang T, Zhu J, George DJ, Armstrong AJ. Enzalutamide versus abiraterone acetate for the treatment of men with metastatic castration-resistant prostate cancer. Expert Opin Pharmacother. 2015 Mar;16(4):473-85. doi: 10.1517/14656566.2015.995090. Epub 2014 Dec 23. PMID 25534660
- [Background] Roubaud G, Liaw BC, Oh WK, Mulholland DJ. Strategies to avoid treatment-induced lineage crisis in advanced prostate cancer. Nat Rev Clin Oncol. 2017 May;14(5):269-283. doi: 10.1038/nrclinonc.2016.181. Epub 2016 Nov 22. PMID 27874061
- [Background] Donkor MK, Sarkar A, Savage PA, Franklin RA, Johnson LK, Jungbluth AA, Allison JP, Li MO. T cell surveillance of oncogene-induced prostate cancer is impeded by T cell-derived TGF-beta1 cytokine. Immunity. 2011 Jul 22;35(1):123-34. doi: 10.1016/j.immuni.2011.04.019. Epub 2011 Jul 14. PMID 21757379
- [Background] Kantoff PW, Higano CS, Shore ND, Berger ER, Small EJ, Penson DF, Redfern CH, Ferrari AC, Dreicer R, Sims RB, Xu Y, Frohlich MW, Schellhammer PF; IMPACT Study Investigators. Sipuleucel-T immunotherapy for castration-resistant prostate cancer. N Engl J Med. 2010 Jul 29;363(5):411-22. doi: 10.1056/NEJMoa1001294. PMID 20818862
- [Background] Yarchoan M, Johnson BA 3rd, Lutz ER, Laheru DA, Jaffee EM. Targeting neoantigens to augment antitumour immunity. Nat Rev Cancer. 2017 Apr;17(4):209-222. doi: 10.1038/nrc.2016.154. Epub 2017 Feb 24. PMID 28233802
- [Background] Rodrigues DN, Rescigno P, Liu D, Yuan W, Carreira S, Lambros MB, Seed G, Mateo J, Riisnaes R, Mullane S, Margolis C, Miao D, Miranda S, Dolling D, Clarke M, Bertan C, Crespo M, Boysen G, Ferreira A, Sharp A, Figueiredo I, Keliher D, Aldubayan S, Burke KP, Sumanasuriya S, Fontes MS, Bianchini D, Zafeiriou Z, Mendes LST, Mouw K, Schweizer MT, Pritchard CC, Salipante S, Taplin ME, Beltran H, Rubin MA, Cieslik M, Robinson D, Heath E, Schultz N, Armenia J, Abida W, Scher H, Lord C, D'Andrea A, Sawyers CL, Chinnaiyan AM, Alimonti A, Nelson PS, Drake CG, Van Allen EM, de Bono JS. Immunogenomic analyses associate immunological alterations with mismatch repair defects in prostate cancer. J Clin Invest. 2018 Nov 1;128(11):5185. doi: 10.1172/JCI125184. Epub 2018 Nov 1. No abstract available. PMID 30382943
- [Background] Whiteside TL. The tumor microenvironment and its role in promoting tumor growth. Oncogene. 2008 Oct 6;27(45):5904-12. doi: 10.1038/onc.2008.271. PMID 18836471
- [Background] Idorn M, Kollgaard T, Kongsted P, Sengelov L, Thor Straten P. Correlation between frequencies of blood monocytic myeloid-derived suppressor cells, regulatory T cells and negative prognostic markers in patients with castration-resistant metastatic prostate cancer. Cancer Immunol Immunother. 2014 Nov;63(11):1177-87. doi: 10.1007/s00262-014-1591-2. Epub 2014 Aug 2. PMID 25085000
- [Background] Dai J, Lu Y, Roca H, Keller JM, Zhang J, McCauley LK, Keller ET. Immune mediators in the tumor microenvironment of prostate cancer. Chin J Cancer. 2017 Mar 14;36(1):29. doi: 10.1186/s40880-017-0198-3. PMID 28292326
- [Background] McAllister MJ, Underwood MA, Leung HY, Edwards J. A review on the interactions between the tumor microenvironment and androgen receptor signaling in prostate cancer. Transl Res. 2019 Apr;206:91-106. doi: 10.1016/j.trsl.2018.11.004. Epub 2018 Nov 24. PMID 30528321
- [Background] Shen YC, Ghasemzadeh A, Kochel CM, Nirschl TR, Francica BJ, Lopez-Bujanda ZA, Carrera Haro MA, Tam A, Anders RA, Selby MJ, Korman AJ, Drake CG. Combining intratumoral Treg depletion with androgen deprivation therapy (ADT): preclinical activity in the Myc-CaP model. Prostate Cancer Prostatic Dis. 2018 Apr;21(1):113-125. doi: 10.1038/s41391-017-0013-x. Epub 2017 Dec 4. PMID 29203894
- [Background] Cha HR, Lee JH, Ponnazhagan S. Revisiting Immunotherapy: A Focus on Prostate Cancer. Cancer Res. 2020 Apr 15;80(8):1615-1623. doi: 10.1158/0008-5472.CAN-19-2948. Epub 2020 Feb 17. PMID 32066566
- [Background] Cai T, Santi R, Tamanini I, Galli IC, Perletti G, Bjerklund Johansen TE, Nesi G. Current Knowledge of the Potential Links between Inflammation and Prostate Cancer. Int J Mol Sci. 2019 Aug 6;20(15):3833. doi: 10.3390/ijms20153833. PMID 31390729
- [Background] Handgretinger R, Lang P, Andre MC. Exploitation of natural killer cells for the treatment of acute leukemia. Blood. 2016 Jun 30;127(26):3341-9. doi: 10.1182/blood-2015-12-629055. Epub 2016 May 20. PMID 27207791
- [Background] Smyth MJ, Cretney E, Kelly JM, Westwood JA, Street SE, Yagita H, Takeda K, van Dommelen SL, Degli-Esposti MA, Hayakawa Y. Activation of NK cell cytotoxicity. Mol Immunol. 2005 Feb;42(4):501-10. doi: 10.1016/j.molimm.2004.07.034. PMID 15607806
- [Background] Liu S, Galat V, Galat Y, Lee YKA, Wainwright D, Wu J. NK cell-based cancer immunotherapy: from basic biology to clinical development. J Hematol Oncol. 2021 Jan 6;14(1):7. doi: 10.1186/s13045-020-01014-w. PMID 33407739
- [Background] Roda JM, Parihar R, Magro C, Nuovo GJ, Tridandapani S, Carson WE 3rd. Natural killer cells produce T cell-recruiting chemokines in response to antibody-coated tumor cells. Cancer Res. 2006 Jan 1;66(1):517-26. doi: 10.1158/0008-5472.CAN-05-2429. PMID 16397268
- [Background] Bottcher JP, Bonavita E, Chakravarty P, Blees H, Cabeza-Cabrerizo M, Sammicheli S, Rogers NC, Sahai E, Zelenay S, Reis e Sousa C. NK Cells Stimulate Recruitment of cDC1 into the Tumor Microenvironment Promoting Cancer Immune Control. Cell. 2018 Feb 22;172(5):1022-1037.e14. doi: 10.1016/j.cell.2018.01.004. Epub 2018 Feb 8. PMID 29429633
- [Background] Brehm C, Huenecke S, Quaiser A, Esser R, Bremm M, Kloess S, Soerensen J, Kreyenberg H, Seidl C, Becker PS, Muhl H, Klingebiel T, Bader P, Passweg JR, Schwabe D, Koehl U. IL-2 stimulated but not unstimulated NK cells induce selective disappearance of peripheral blood cells: concomitant results to a phase I/II study. PLoS One. 2011;6(11):e27351. doi: 10.1371/journal.pone.0027351. Epub 2011 Nov 9. PMID 22096557
- [Background] Wu X, Matosevic S. Gene-edited and CAR-NK cells: Opportunities and challenges with engineering of NK cells for immunotherapy. Mol Ther Oncolytics. 2022 Nov 3;27:224-238. doi: 10.1016/j.omto.2022.10.011. eCollection 2022 Dec 15. PMID 36420307
- [Background] Sakamoto N, Ishikawa T, Kokura S, Okayama T, Oka K, Ideno M, Sakai F, Kato A, Tanabe M, Enoki T, Mineno J, Naito Y, Itoh Y, Yoshikawa T. Phase I clinical trial of autologous NK cell therapy using novel expansion method in patients with advanced digestive cancer. J Transl Med. 2015 Aug 25;13:277. doi: 10.1186/s12967-015-0632-8. PMID 26303618
- [Background] Miller JS, Soignier Y, Panoskaltsis-Mortari A, McNearney SA, Yun GH, Fautsch SK, McKenna D, Le C, Defor TE, Burns LJ, Orchard PJ, Blazar BR, Wagner JE, Slungaard A, Weisdorf DJ, Okazaki IJ, McGlave PB. Successful adoptive transfer and in vivo expansion of human haploidentical NK cells in patients with cancer. Blood. 2005 Apr 15;105(8):3051-7. doi: 10.1182/blood-2004-07-2974. Epub 2005 Jan 4. PMID 15632206
- [Background] Rubnitz JE, Inaba H, Ribeiro RC, Pounds S, Rooney B, Bell T, Pui CH, Leung W. NKAML: a pilot study to determine the safety and feasibility of haploidentical natural killer cell transplantation in childhood acute myeloid leukemia. J Clin Oncol. 2010 Feb 20;28(6):955-9. doi: 10.1200/JCO.2009.24.4590. Epub 2010 Jan 19. PMID 20085940
- [Background] Iliopoulou EG, Kountourakis P, Karamouzis MV, Doufexis D, Ardavanis A, Baxevanis CN, Rigatos G, Papamichail M, Perez SA. A phase I trial of adoptive transfer of allogeneic natural killer cells in patients with advanced non-small cell lung cancer. Cancer Immunol Immunother. 2010 Dec;59(12):1781-9. doi: 10.1007/s00262-010-0904-3. Epub 2010 Aug 12. PMID 20703455
- [Background] Scher HI, Morris MJ, Stadler WM, Higano C, Basch E, Fizazi K, Antonarakis ES, Beer TM, Carducci MA, Chi KN, Corn PG, de Bono JS, Dreicer R, George DJ, Heath EI, Hussain M, Kelly WK, Liu G, Logothetis C, Nanus D, Stein MN, Rathkopf DE, Slovin SF, Ryan CJ, Sartor O, Small EJ, Smith MR, Sternberg CN, Taplin ME, Wilding G, Nelson PS, Schwartz LH, Halabi S, Kantoff PW, Armstrong AJ; Prostate Cancer Clinical Trials Working Group 3. Trial Design and Objectives for Castration-Resistant Prostate Cancer: Updated Recommendations From the Prostate Cancer Clinical Trials Working Group 3. J Clin Oncol. 2016 Apr 20;34(12):1402-18. doi: 10.1200/JCO.2015.64.2702. Epub 2016 Feb 22. PMID 26903579
- [Background] Barbosa FG, Queiroz MA, Ferraro DA, Nunes RF, Dreyer PR, Zaniboni EC, Costa LB, Bastos DA, Marin JFG, Buchpiguel CA. Prostate-specific Membrane Antigen PET: Therapy Response Assessment in Metastatic Prostate Cancer. Radiographics. 2020 Sep-Oct;40(5):1412-1430. doi: 10.1148/rg.2020200058. Epub 2020 Aug 7. PMID 32762625
- [Background] Yuan Y, Hess KR, Hilsenbeck SG, Gilbert MR. Bayesian Optimal Interval Design: A Simple and Well-Performing Design for Phase I Oncology Trials. Clin Cancer Res. 2016 Sep 1;22(17):4291-301. doi: 10.1158/1078-0432.CCR-16-0592. Epub 2016 Jul 12. PMID 27407096
- [Background] Lee DW, Santomasso BD, Locke FL, Ghobadi A, Turtle CJ, Brudno JN, Maus MV, Park JH, Mead E, Pavletic S, Go WY, Eldjerou L, Gardner RA, Frey N, Curran KJ, Peggs K, Pasquini M, DiPersio JF, van den Brink MRM, Komanduri KV, Grupp SA, Neelapu SS. ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells. Biol Blood Marrow Transplant. 2019 Apr;25(4):625-638. doi: 10.1016/j.bbmt.2018.12.758. Epub 2018 Dec 25. PMID 30592986
- [Background] Kottaridis PD, North J, Tsirogianni M, Marden C, Samuel ER, Jide-Banwo S, Grace S, Lowdell MW. Two-Stage Priming of Allogeneic Natural Killer Cells for the Treatment of Patients with Acute Myeloid Leukemia: A Phase I Trial. PLoS One. 2015 Jun 10;10(6):e0123416. doi: 10.1371/journal.pone.0123416. eCollection 2015. PMID 26062124
- [Background] Fehniger TA, Miller JS, Stuart RK, Cooley S, Salhotra A, Curtsinger J, Westervelt P, DiPersio JF, Hillman TM, Silver N, Szarek M, Gorelik L, Lowdell MW, Rowinsky E. A Phase 1 Trial of CNDO-109-Activated Natural Killer Cells in Patients with High-Risk Acute Myeloid Leukemia. Biol Blood Marrow Transplant. 2018 Aug;24(8):1581-1589. doi: 10.1016/j.bbmt.2018.03.019. Epub 2018 Mar 27. PMID 29597002
- [Background] Lowdell MW, Craston R, Samuel D, Wood ME, O'Neill E, Saha V, Prentice HG. Evidence that continued remission in patients treated for acute leukaemia is dependent upon autologous natural killer cells. Br J Haematol. 2002 Jun;117(4):821-7. doi: 10.1046/j.1365-2141.2002.03495.x. PMID 12060116
- See also: Tracy, C. (2022). Prostate Cancer Treatment & Management: Approach Considerations, Localized Prostate Cancer, Management of Advanced and Metastatic Disease. — http://emedicine.medscape.com/article/1967731-treatment
- See also: FDA (2021). Drug Development Tools: Fit-for-Purpose Initiative — http://www.fda.gov/drugs/development-approval-process-drugs/drug-development-tools-fit-purpose-initiative